CLINICAL TRIAL: NCT03789045
Title: New Methodological Approach to Metabolic Thresholds Detection; Examining Fat Utilization Points and Metabolic Thresholds Correlation Strength
Brief Title: Metabolic Thresholds and Fat Utilization Points Correlation
Acronym: MATDFP
Status: Completed | Type: Observational
Sponsor: Sport Studio Banja Luka (Other)
Collaborators: Aspire Medical (Industry); Appalachian State University (Other); University of South Australia (Other); University Ghent (Other); University of Birmingham (Other); Stanford University (Other); Cosmed USA, Inc. (Industry); University Hospital of Split (Other); University of Urbino "Carlo Bo" (Other); Universidad de Granada (Other); Autonomous University of Ciudad Juarez (Unknown)
Responsible Party: Principal Investigator, Ratko Peric, Exercise Physiologist PhD, Sport Studio Banja Luka
Other Study IDs: 12345
Record Dates: First submitted 2018-12-21; First posted 2018-12-28 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Exercise Physiology
Keywords: Exercise; Metabolic thresholds; Fat oxidation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Obese men and women: Metabolic thresholds and fat oxidation points relationship in Obese males and females, age 18-60y, body fat > 30%
  Interventions: Diagnostic Test: Metabolic thresholds and fat oxidation points relationship
- Male and female athletes: Metabolic thresholds and fat oxidation points relationship in Athletic males and females, age 18-60y.
  Interventions: Diagnostic Test: Metabolic thresholds and fat oxidation points relationship
- Sedentary females and males: Metabolic thresholds and fat oxidation points relationship in Sedentary females and males, age 18-60y,
  Interventions: Diagnostic Test: Metabolic thresholds and fat oxidation points relationship

INTERVENTIONS:
Diagnostic Test: Metabolic thresholds and fat oxidation points relationship — Investigators aim to determine exercise intensity at which metabolic thresholds and fat oxidation points occur by using non-invasive breath-by-breath gas analysis during either graded treadmill or cycle ergometry test (2min stages and 1km/h or 50 W load increase) till exhaustion to determine maximal oxygen uptake (VO2max), with gases being collected at the mouth level. The strength of the relationship between AeT and at FATmax will be assessed using the Pearson product moment (r) correlation coefficient with same being done for AnT and FATmin correlation. A coefficient of determination (R2) will be used to detect the proportion of existing variance. A paired t-test will be used to asses' differences between measured variables. Bland-altman will be used to determine levels of agreement.

SUMMARY:
To examine existence of connection between fat utilization points, both maximal and minimal with individual metabolic thresholds in different subjects. As a consequence, this innovative approach could offer a supplementary method for both aerobic and anaerobic thresholds detection as well as useful and practical exercise intensity selection marker.

DETAILED DESCRIPTION:
This study aims to examine the existence of connection between metabolic thresholds and fat oxidation points in diverse group of subjects. From the physiological perspective, during exercise with increasing intensity, three phases of the body's energy utilization and two threshold points can be defined. These threshold points have been named metabolic thresholds and as such are considered as indicators of exercise capacities. Several authors have suggested, that the first threshold should be called the 'aerobic threshold' (AeT) and the second the 'anaerobic threshold' (AnT). The energy contribution from fat oxidation increases during low-to-moderate exercise intensities and then markedly declines when the intensity becomes high, at which point carbohydrates (CHO) remain the dominant energy substrate. A term used to describe exercise intensity where fat oxidation reaches optimum, is maximal fat oxidation point (FATmax) whereas exercise intensity matching the negligible fat oxidation is labelled FATmin. During physical activity, due to limited availability of CHO, subjects are more dependent on energy originating from fat when aiming to optimize endurance performance, body composition, optimize weight control and the metabolic rate. Exercise at the intensity eliciting FATmax revealed best results in treatment and prevention of obesity-associated conditions, cardio-vascular and pulmonary diseases by means of increase in maximal fat oxidation rates (MFO), insulin sensitivity, improvements in ventilator efficiency and cardiac output, demonstrating a significant role in the treatment of these impairments. As a follow-up, studies demonstrated how the lowest beneficial effect was observed when exercise was performed above intensity matching negligible fat oxidation rate (FATmin), contributing to diminished protection of exercise therapy. In consequence, increased cardio-metabolic demands of exercise performed above FATmin also have a higher impact on mortality rates in comparison to low-moderate aerobic exercise. Therefore, choosing appropriate exercise intensity may play a decisive role in decreasing risk factors accompanying obesity-associated conditions.

Investigators aim to determine metabolic thresholds and fat oxidation points by using non-invasive breath-by-breath gas analysis during either treadmill or cycle ergometry. Metabolic thresholds will be detected by using gas analysis, via ventilatory parameters. Fat oxidation points will be determined using indirect calorimetry.

Participants will perform graded ergometry test (2min stages and 1km/h or 50 W load increase), on either cycle or treadmill ergometer, till exhaustion to determine maximal oxygen uptake (VO2max), with gases being collected at the mouth level by using spiroergometry.

The strength of the relationship between intensities matching VO2 at AeT and VO2 at FATmax will be assessed using the Pearson product moment (r) correlation coefficient with same being done for AnT and FATmin correlation. A coefficient of determination (R2) will be used to detect the proportion of existing variance. A paired t-test will be used to asses' differences between measured variables.

Associated heart rate at the AeT/FATmax and AnT/FATmin will be used as training mean to identify proper training intensity.

The time frame of the study is about 3 years, depending on the availability of the subjects. Planed study begin is early 2016. Participants will be every day clients of the Institution and will be recruited on a voluntary basis as they arrive to the testing facilities through this 3 years period.Through this 3 years period, statistical analysis of the collected data for each group of subjects will be performed and observations will be published. Up to 7 publications are expected to result from this research.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non smokers
* No evidence of any metabolic, pulmonary or cardiovascular diseases possibly affecting substrates utilization.
* No presence of musculoskeletal injuries (Must be able to perform graded exercise test on a treadmill or a cycle ergometer).
* Males and females, age 18-60, divided in following 4 groups: obese, sedentary, moderately trained, athletes.
* For obese group of individuals, body fat > 30%
* For sedentary group of individuals, no physical activity in last 3 years
* For athletic group of individuals, > 12 h training per week
* For moderately trained individuals. < 3 h per week of physical activity
* Willing to allow data publication.

Exclusion Criteria:

* Evidence of any metabolic, pulmonary or cardiovascular diseases possibly affecting substrates utilization.
* Smokers.
* High blood pressure.
* Using supplements possibly affecting substrates utilization.
* Non willing to allow data publication.
* Not finishing grade exercise test protocol till exhaustion to determine VO2max.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Athletic, moderately trained, sedentary and obese males and females
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Relationship between metabolic threshold and fat oxidation points (FATmax) matching %HRmax | Each primary outcome measure (metabolic thresholds and fat oxidation points, is sampled continuously through the test. Test duration is 12-16 minutes.Existence of correlation will be evaluated immediately after test
  Regular exercise at FATmax intensity has been proposed as a key factor to optimize the body's ability to oxidize lipids.Exercise intensity matching FATmax will be determined via indirect calorimetry and expressed by using %HRmax.In contrast to the %HRmax method, an individualized approach to exercise intensity prescription based on metabolic thresholds describes specific metabolic phases during exercise and intends to account for differences in the body's physiological and functional capacity.Metabolic thresholds will be determined via either gas analysis or/and lactate analysis and expressed in %HRmax.If connection between these two %HRmax exists,it would integrate the most relevant indices for planning and assessing an effective exercise program.Existence of connection between %HRmax matching both parameters will be evaluated by using correlation and levels of agreement by using MedCalc statistical software.

SECONDARY OUTCOMES:
Relationship between metabolic threshold and fat oxidation points (FATmax) matching %VO2max | Each primary outcome measure (metabolic thresholds and fat oxidation points, is sampled continuously through the test. Test duration is 12-16 minutes. Existence of correlation will be evaluated immediately after test
  Regular exercise at FATmax intensity has been proposed as a key factor to optimize the body's ability to oxidize lipids.Exercise intensity matching FATmax will be determined via indirect calorimetry and expressed by using %VO2max.In contrast to the %VO2max method, an individualized approach to exercise intensity prescription based on metabolic thresholds describes specific metabolic phases during exercise and intends to account for differences in the body's physiological and functional capacity.Metabolic thresholds will be determined via either gas analysis or/and lactate analysis and expressed in %VO2max.If connection between these two %VO2max exists, it would integrate the most relevant indices for planning and assessing an effective exercise program.Existence of connection between %VO2max matching both parameters will be evaluated by using correlation and levels of agreement by using MedCalc statistical software.

CONTACTS AND LOCATIONS:
Overall Officials: Ratko Peric, Doctorate, Principal Investigator — Sport Studio Banja Luka
Locations (1):
- Sport Studio Banja Luka, Banja Luka, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be made available upon request. Raw sampling data or statistical analysis data

REFERENCES:
- [Background] Peric R, DI Pietro A, Myers J, Nikolovski Z. A systematic comparison of commonly used stoichiometric equations to estimate fat oxidation during exercise in athletes. J Sports Med Phys Fitness. 2021 Oct;61(10):1354-1361. doi: 10.23736/S0022-4707.20.11747-X. Epub 2020 Dec 14. PMID 33314884
- [Result] Peric R, Meucci M, Nikolovski Z. Fat Utilization During High-Intensity Exercise: When Does It End? Sports Med Open. 2016 Dec;2(1):35. doi: 10.1186/s40798-016-0060-1. Epub 2016 Aug 31. PMID 27747790
- [Result] Peric R, Meucci M, Bourdon PC, Nikolovski Z. Does the aerobic threshold correlate with the maximal fat oxidation rate in short stage treadmill tests? J Sports Med Phys Fitness. 2018 Oct;58(10):1412-1417. doi: 10.23736/S0022-4707.17.07555-7. Epub 2017 Jul 25. PMID 28745473
- [Result] Meucci M, Peric R. Correlation Between Aerobic Threshold And Point Of Maximal Fat Utilization In Male Runners: 1678 Board #331 June 2, 8: 00 AM - 9: 30 AM. Med Sci Sports Exerc. 2016 May;48(5 Suppl 1):466-7. doi: 10.1249/01.mss.0000486403.83644.7e.
- [Result] Peric R, Nikolovski Z. Can metabolic thresholds be used as exercise intensity markers in adult men with obesity - fat burn points used as an exercise marker. Comparative Exercise Physiology: 16 (2)- Pages: 113 - 119. https://doi.org/10.3920/CEP190035
- [Result] Nikolovski Z, Barbaresi S, Cable T, Peric R. Evaluating the influence of differences in methodological approach on metabolic thresholds and fat oxidation points relationship. Eur J Sport Sci. 2021 Jan;21(1):61-68. doi: 10.1080/17461391.2020.1717640. Epub 2020 Jan 31. PMID 31944160
- [Result] Meucci M, Nandagiri V, Kavirayuni VS, Whang A, Collier SR. Correlation Between Heart Rate at Maximal Fat Oxidation and Aerobic Threshold in Healthy Adolescent Boys and Girls. Pediatr Exerc Sci. 2021 May 6;33(3):139-143. doi: 10.1123/pes.2020-0210. PMID 33958504
- [Result] Peric R, Nikolovski Z, Meucci M, Tadger P, Ferri Marini C, Amaro-Gahete FJ. A Systematic Review and Meta-Analysis on the Association and Differences between Aerobic Threshold and Point of Optimal Fat Oxidation. Int J Environ Res Public Health. 2022 May 26;19(11):6479. doi: 10.3390/ijerph19116479. PMID 35682065
- [Result] Ferri Marini C, Tadger P, Chavez-Guevara IA, Tipton E, Meucci M, Nikolovski Z, Amaro-Gahete FJ, Peric R. Factors Determining the Agreement between Aerobic Threshold and Point of Maximal Fat Oxidation: Follow-Up on a Systematic Review and Meta-Analysis on Association. Int J Environ Res Public Health. 2022 Dec 27;20(1):453. doi: 10.3390/ijerph20010453. PMID 36612784